CLINICAL TRIAL: NCT06370286
Title: The Effect of Acute Concurrent Exercise on Inhibitory Control: An Event-related Potential Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACNL_rueihongli_CE_IC
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Exercise; Cognition
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either a concurrent exercise (CE), aerobic exercise (AE), or control (CON) group. Participants in the CE group engaged in 12-minutes of AE (40%-59% of heart rate reserve [HRR]) coupled with 13-minutes of resistance exercise (1 set, with 75% of 10-repetition maximum, and 12 repetitions of 8 movements). The AE group participated in 25 minutes of AE (40%-59% HRR). Prior to and following exercise onset, participants in both the CE and AE groups completed a 5-minute warm-up and cool-down. Participants in the CON group read books for 35 minutes. Lactate concentrations were measured at timepoint of 0-, 17-, and 30-minutes relative to the treatment onset. Response time (RT) and accuracy in the Stroop test, as well as P3 amplitudes, were assessed before and after the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- concurrent exercise (CE) (Experimental): Participants in the concurrent exercise group engaged in 12-minutes of aerobic exercise (40%-59% of heart rate reserve [HRR]) coupled with 13-minutes of resistance exercise (1 set, with 75% of 10-repetition maximum, and 12 repetitions of 8 movements). Prior to and following exercise onset, participants completed a 5-minute warm-up and cool-down.
  Interventions: Behavioral: concurrent exercise (CE)
- aerobic exercise (AE) (Experimental): Participants in the aerobic exercise (AE) group participated in 25 minutes of AE (40%-59% of heart rate reserve [HRR]). Prior to and following exercise onset, participants completed a 5-minute warm-up and cool-down.
  Interventions: Behavioral: aerobic exercise (AE)
- control (CON) (No Intervention): Participants in the control group read books for 35 minutes.

INTERVENTIONS:
Behavioral: concurrent exercise (CE) — Participants in the concurrent exercise group engaged in 12-minutes of aerobic exercise (40%-59% of heart rate reserve [HRR]) coupled with 13-minutes of resistance exercise (1 set, with 75% of 10-repetition maximum, and 12 repetitions of 8 movements). Prior to and following exercise onset, participants completed a 5-minute warm-up and cool-down.
  Arms: concurrent exercise (CE)
Behavioral: aerobic exercise (AE) — Participants in the aerobic exercise (AE) group participated in 25 minutes of AE (40%-59% of heart rate reserve [HRR]). Prior to and following exercise onset, participants completed a 5-minute warm-up and cool-down.
  Arms: aerobic exercise (AE)

SUMMARY:
The present study aimed to determine the effects of acute concurrent exercise on inhibitory control via behavioral and event-related potential approaches and to examine its potential mediational role on lactate among younger adults. The main questions it aims to answer are: (1) Does acute concurrent exercise improve inhibitory control via behavioral and event-related potential approaches? (2) Does lactate play a potential mediational role in the effect of acute concurrent exercise on inhibitory control?

DETAILED DESCRIPTION:
The present study aimed to determine the effects of acute concurrent exercise (CE) on inhibitory control via behavioral and event-related potential approaches and to examine its potential mediational role on lactate. Participants were randomly assigned to either a CE, aerobic exercise (AE), or control (CON) group. Participants in the CE group engaged in 12-minutes of AE (40%-59% of heart rate reserve [HRR]) coupled with 13-minutes of resistance exercise (1 set, with 75% of 10-repetition maximum, and 12 repetitions of 8 movements). The AE group participated in 25 minutes of AE (40%-59% HRR). Prior to and following exercise onset, participants in both the CE and AE groups completed a 5-minute warm-up and cool-down. Participants in the CON group read books for 35 minutes. Lactate concentrations were measured at timepoint of 0-, 17-, and 30-minutes relative to the treatment onset. Response time (RT) and accuracy in the Stroop test, as well as P3 amplitudes, were assessed before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 30 years
* able to exercise without undue risk (i.e., the first seven questions of the Physical Activity Readiness Questionnaire for Everyone [PAR-Q+] were answered "No")
* right-handed dominance
* typical or corrected-to-typical eyesight
* limited physical activity in the previous month (i.e., < 150 minutes/week of moderate-intensity physical activity)

Exclusion Criteria:

* psychiatric or neurological ailments
* cardiorespiratory or neuromuscular conditions
* obese status (body mass index [BMI] > 27 kg/m2)

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 78 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Inhibitory control | 30 minutes
  Inhibitory control was assessed using a modified computerized version of the Stroop test, which was administered through Neuroscan Stim2 software (Compumedics Neuroscan, Charlotte, NC). The test comprised four blocks, each consisting of 108 trials. Within each block, three types of trials were presented: neutral, congruent, and incongruent. The neutral trial involved displaying a square printed in red, green, or blue color. The congruent trial presented Chinese language prints in corresponding colors and words [i.e., 紅 (RED), 綠 (GREEN), or 藍 (BLUE)]. In contrast, the incongruent trial displayed Chinese language prints in different colors and words [e.g., 紅 (RED) printed in blue color]. Each block included 36 neutral trials, 36 congruent trials, and 36 incongruent trials. Participants were instructed to respond promptly and accurately to the color of the stimulus presented. Subsequently, the mean response time (RT) of correct trials and accuracy for each Stroop condition were examined.

SECONDARY OUTCOMES:
Blood lactate | Timepoint 1 (prior to the commencement of treatment), Timepoint 2 (17 minutes after the initiation of treatment), and Timepoint 3 (30 minutes after the start of treatment).
  Blood lactate levels were assessed using fingertip samples measured with a lactate analyzer (The EDGE, Taipei, Taiwan) at three distinct time points: Timepoint 1 (prior to the commencement of treatment), Timepoint 2 (17 minutes after the initiation of treatment), and Timepoint 3 (30 minutes after the start of treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, PhD, Study Chair — Department of Physical Education and Sport Sciences, National Taiwan Normal University; Ruei-Hong Li, MS, Principal Investigator — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (1):
- Department of Physical Education and Sport Sciences, National Taiwan Normal University, Taipei, Taiwan

REFERENCES:
- [Derived] Li RH, Chen TR, Gilson ND, Brazaitis M, Cheng YT, Wu HF, Lee JH, Chang YK. Acute Concurrent Exercise Improves Inhibitory Control Without Mediating the Role of Lactate: An Event-Related Potential Study. Sports Med Open. 2025 Jan 27;11(1):12. doi: 10.1186/s40798-024-00809-2. PMID 39871026